CLINICAL TRIAL: NCT05482269
Title: Prediction of Adverse Outcome of Acute Pulmonary Embolism by Artificial Intelligence System Based on CT Pulmonary Angiography
Brief Title: Adverse Outcome of Acute Pulmonary Embolism by Artificial Intelligence System Based on CT Pulmonary Angiography
Acronym: PEAICTPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, YIZHUO GAO, Doctor, Shengjing Hospital
Other Study IDs: PEAICTPA
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Embolism and Thrombosis; Deterioration, Clinical; Artificial Intelligence
Keywords: Pulmonary Embolism and Thrombosis; Deterioration, Clinical; Artificial Intelligence
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis; Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The investigators aim to build a predictive tool for Adverse Outcome of Acute Pulmonary Embolism by Artificial Intelligence System Based on CT Pulmonary Angiography.

DETAILED DESCRIPTION:
This study collected clinical, laboratory, and CT parameters of acute patients with acute pulmonary embolism from admission to predict adverse outcomes within 30 days after admission into hospital. The investigators aim to build a predictive tool for Adverse Outcome of Acute Pulmonary Embolism by Artificial Intelligence System Based on CT Pulmonary Angiography.

Eligible patients were randomized in some ratio into derivation and validation cohorts. The derivation cohort was used to develop and evaluate a multivariable logistic regression model for predicting the outcomes of interest. The discriminatory power was evaluated by comparing the nomogram to the established risk stratification systems. The consistency of the nomogram was evaluated using the validation cohort.

ELIGIBILITY:
Inclusion Criteria:

* age of ≥ 18 years and a pulmonary embolism diagnosis based on CT pulmonary angiography

Exclusion Criteria:

* pregnancy
* reception of reperfusion treatment before admission
* missing data regarding CT parameters, echocardiography, cardiac troponin I (c-Tn I), and N-terminal-pro brain natriuretic peptide (NT-pro BNP) levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 30 days
  The outcomes of interest were defined as the occurrence of adverse outcomes within 30 days after admission. Adverse outcomes were defined as deaths, the need for mechanical ventilation, the need for cardiopulmonary resuscitation, and the need for life-saving vasopressor and reperfusion treatment.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years
  The outcomes of interest were defined as the occurrence of adverse outcomes within 2 years after admission. Adverse outcomes were defined as deaths, the need for mechanical ventilation, the need for cardiopulmonary resuscitation, and the need for life-saving vasopressor and reperfusion treatment.

CONTACTS AND LOCATIONS:
Overall Officials: DONG JIA, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided